CLINICAL TRIAL: NCT03162419
Title: To Assess the Efficacy of High-Volume Plasma Exchange and GCSF Versus GCSF Alone in Patients of Acute on Chronic Liver Failure (ACLF)-A Randomized Controlled Trial.
Brief Title: To Assess the Efficacy of High-Volume Plasma Exchange and GCSF Versus GCSF Alone in Patients of Acute on Chronic Liver Failure (ACLF).
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Funds.
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ACLF-01
Record Dates: First submitted 2017-04-20; First posted 2017-05-22 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-06

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Plasma Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Medical Therapy (Active Comparator): The patients in group A will be given standard medical therapy only as per requirement. Lactulose, bowel wash, albumin, terlipressin, antibiotics and anti-virals in hepatitis B reactivation will be continued and recorded.
  Interventions: Drug: Standard Medical Therapy
- Standard Medical Therapy + Plasma exchange + GCSF (Experimental): The patients in group B shall be given GCSF in a dose of 5 ug/kg/day on day 1,2,3,4,5 followed by every 3rd day till day 28 along with alternate day high volume plasma exchange sessions till a maximum of ten sessions.
  Interventions: Drug: Standard Medical Therapy; Biological: Plasma Exchange; Biological: GCSF
- Standard Medical Therapy + GCSF (Experimental): The patients in this will be given standard medical therapy only as per requirement. Lactulose, bowel wash, albumin, terlipressin, antibiotics and anti-virals in hepatitis B reactivation will be continued and recorded.
  The GCSF in a dose of 5 ug/kg/day on day 1,2,3,4,5 followed by every 3rd day till day 28
  Interventions: Drug: Standard Medical Therapy; Biological: GCSF

INTERVENTIONS:
Drug: Standard Medical Therapy — The patients in group A will be given standard medical therapy only as per requirement. Lactulose, bowel wash, albumin, terlipressin, antibiotics and anti-virals in hepatitis B reactivation will be continued and recorded.
Biological: Plasma Exchange — High volume plasma exchange sessions till a maximum of ten sessions.
  Arms: Standard Medical Therapy + Plasma exchange + GCSF
Biological: GCSF — The GCSF in a dose of 5 ug/kg/day on day 1,2,3,4,5 followed by every 3rd day till day 28
  Arms: Standard Medical Therapy + GCSF; Standard Medical Therapy + Plasma exchange + GCSF

SUMMARY:
Study design-Open label randomized controlled trial

Study period-2 years

Study population-All patients of ACLF admitted to ILBS for a period of two years from Feb 2017 to Dec 2018

All the patients of ACLF will receive standard medical therapy and will be randomized within 48 hours of admission into three groups after screening for exclusion and inclusion criteria.(1:2:2) Group A-Standard Medical Therapy only Group B-Standard Medical therapy + Plasma exchange + GCSF Group C-Standard Medical Therapy + GCSF

ELIGIBILITY:
Inclusion Criteria:

- All consecutive patients in age group of 18-70 years with acute on chronic liver failure as defined by APASL criteria shall be included in the study.Only those patients who wish to be enrolled in the trial shall be included in the study.

Exclusion Criteria:

1. Steroid eligible patients with severe alcoholic hepatitis
2. Cirrhosis of liver with previous history of decompensation
3. Patients with severe cardiopulmonary disease
4. Pregnancy
5. Human Immmunodeficiency Virus infection
6. Hepatocellular carcinoma or extrahepatic malignancy
7. Chronic renal insufficiency on treatment with haemodialysis
8. Uncontrolled bleed or patients in disseminated intravascular coagulopathy
9. Patient with expected survival of less than 48 hours
10. Patients with moderate-severe acute respiratory distress syndrome
11. Hemodynamic instability with noradrenaline requirement of more than >0.5ug/kg/min or requirement of dual vasopressors
12. Patients with leukemoid reaction or total leucocyte count > 40,000/mm3
13. Patients diagnosed with Hemophagocytic Lymphohistiocytosis
14. Patients with known hypersensitivity to Granulocyte colony stimulating factor

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-04-25 (Estimated); Study Completion 2019-04-25 (Estimated)

PRIMARY OUTCOMES:
Transplant free survival | 28 days

SECONDARY OUTCOMES:
Improvement in biochemical parameter which is defined as > 20% reduction from baseline in both groups | Day 14
Improvement in biochemical parameter which is defined as > 20% reduction from baseline in both groups | Day 28
Improvement in clinical parameters which is defined as > 20% reduction from baseline in both groups | Day 14
Improvement in clinical parameters which is defined as > 20% reduction from baseline in both groups | Day 28
Improvement in APACHEII (by 2 points ) | 2 years
Improvement in MELD (by 2 points ) | 2 years
Improvement in SIRS by 2 points | 2 years
Improvement in SOFA (by 2 points ) | 2 years
Incidence of new onset sepsis and SIRS in both groups. | Day 28
Side effects of therapy in both groups | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No